CLINICAL TRIAL: NCT06693063
Title: Impact of General Practice Follow-up on Emergency Hospitalization of Patients Admitted for Chest Pain
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor
Other Study IDs: EDS_2024_douleurthoracique
Record Dates: First submitted 2024-11-08; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Chest Pain
Keywords: emergency admission; general practitioner
MeSH Terms: conditions — Chest Pain | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient followed by a general practitionner: GP consulted in the last 12 months
  Interventions: Other: Data collection
- Patient not followed by a general practitionner: Patient without regular follow-up
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Some data will be collected for all patients included: medical and family history, chest pain data and medical care data

SUMMARY:
This is a prospective observational study carried out in the emergency department of Emile Roux Hospital. Its aim is to compare the medical, psychological and social characteristics of patients followed up by a general practitioner and those without regular follow-up, using an anonymous questionnaire completed by the general practitioner in the emergency department, for patients consulting for the reason "chest pain".

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to Emile Roux hospital emergency department with chest pain
* Patient affiliated to the Social security system
* Patient able to give informed non-opposition to participating in research

Exclusion Criteria:

* Patient under guardianship, curatorship, safeguard of justice or prisoners
* Patient with cognitive disorders
* Pregnant or breast-feeding women
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to Emile Roux hospital emergency department with chest pain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Compare the hospitalization rate of patients admitted for chest pain, according to their medical follow-up by a general practitioner. | Only once, within 24 hours of admission to the emergency department

SECONDARY OUTCOMES:
Describe the population of patients admitted to the Emile Roux hospital emergency department with chest pain and followed by a general practitioner versus those without medical follow-up. | Only once, within 24 hours of admission to the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Luc PIGEON, Principal Investigator — Hospital Center Emile Roux, Le Puy-en-Velay (France)
Locations (1):
- Centre Hospitalier Emile Roux, Le Puy-en-Velay, France

IPD SHARING:
Plan to Share IPD: Undecided